CLINICAL TRIAL: NCT06060691
Title: Randomized Controlled Trial Studying the Ameliorating Effects of Kaempferol Emulgel on Female Arousal Disorder and Sexual Dysfunction
Brief Title: the Ameliorating Effects of Antioxidant Gel on Female Arousal Disorder and Sexual Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5/23
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Female Sexual Dysfunction
MeSH Terms: interventions — kaempferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kaempferol group (Experimental): Kaempferol gel received the vaginal gel containing antioxidant extract every day for seven days. Then, the treatment continued for two months, twice weekly
  Interventions: Drug: Kaempferol
- Placebo group (Placebo Comparator): Plain formulation received the vaginal gel containing antioxidant extract every day for seven days. Then, the treatment continued for two months, twice weekly
  Interventions: Drug: Kaempferol

INTERVENTIONS:
Drug: Kaempferol — Kaempferol

SUMMARY:
The aim of this study is to evaluate the quality of sexual life of females with sexual interest or arousal disorder before and after accurate application of a formulated emulgel made from natural ingredients, including kaempferol as an API

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 28 and 45
* had regular periods and previous menstrual bleeding lasted between three and seven days

Exclusion Criteria:

* sensitivity to drug of therapy,
* cancer,
* autoimmune illness,
* smoking or drinking,
* liver disease,
* irregular menstruation

Ages: 28 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female has sexual problems
Enrollment: 30 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index | two months
  The FSFI comprises 19 questions of sexual function in six independent areas consisting of desire, arousal, lubrication, orgasm, sexual satisfaction , pain from sex.

CONTACTS AND LOCATIONS:
Locations (1):
- Soad A. Mohamad, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No